CLINICAL TRIAL: NCT02235662
Title: Phase I One-Month Safety, Pharmacokinetic, Pharmacodynamic, and Acceptability Study of Intravaginal Rings Releasing Tenofovir and Levonorgestrel or Tenofovir Alone
Brief Title: Phase I One-month Safety, PK, PD, and Acceptability Study of IVR Releasing TFV and LNG or TFV Alone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A13-128
Record Dates: First submitted 2014-07-14; First posted 2014-09-10 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: HIV; Contraception
Keywords: HIV; LNG; IVR; Contraception; Prevention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TFV IVR (Experimental): TFV IVR is an intravaginal ring 55.0 mm in diameter, consisting of single segment of polyurethane tubing with an outer diameter of 5.5 mm and filled with white TFV-containing paste. Used for one month, the IVR delivers 8-10 mg/day TFV.
  Interventions: Drug: TFV IVR
- TFV/LNG IVR (Experimental): TFV/LNG IVR is an intravaginal ring 55.0 mm in diameter, consisting of two segments of polyurethane tubing with an outer diameter of 5.5 mm: a longer segment containing white TFV paste and a shorter one (20 mm) with a white LNG core. Used for one month, the IVR delivers 8-10 mg/day TFV and 20 μg/day LNG.
  Interventions: Drug: TFV IVR; Drug: TFV/LNG IVR
- Placebo Intravaginal Ring (Placebo Comparator): Intravaginal ring 55.0 mm in diameter, consisting of two segments of polyurethane tubing with an outer diameter of 5.5 mm containing no active experimental ingredients. Used for one month.
  Interventions: Other: Placebo IVR

INTERVENTIONS:
Drug: TFV IVR
  Other Names: Tenofovir Intravaginal Ring
  Arms: TFV IVR; TFV/LNG IVR
Drug: TFV/LNG IVR
  Other Names: Tenofovir Levonorgestrel Intravaginal Ring
  Arms: TFV/LNG IVR
Other: Placebo IVR
  Other Names: Placebo Intravaginal Ring
  Arms: Placebo Intravaginal Ring

SUMMARY:
The purpose of the study is to evaluate the safety of the TFV/LNG intravaginal ring (IVR), TFV-only IVR, and placebo IVR, evaluate pharmacokinetics (PK) of TFV and LNG, evaluate pharmacodynamic (PD) surrogates of contraceptive efficacy of LNG, and to evaluate acceptability of the IVRs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years, inclusive
* General good health (by volunteer history and per investigator discretion) without any clinically significant systemic disease (including, but not limited to significant liver disease/hepatitis, gastrointestinal disease, kidney disease, thyroid disease, osteoporosis or bone disease, and diabetes)
* Currently having regular menstrual cycles of 26-35 days by participant report
* History of Pap smears and follow-up consistent with standard medical practice as outlined in the study manual or willing to undergo a Pap smear
* Protected from pregnancy by one of the following: 1) Sterilization of either partner. Note: Women protected from pregnancy by sterilization of either partner must abstain from vaginal intercourse from 48 hours prior to Visit 3 until the sixth day after the last study visit; or 2) Willing to abstain from vaginal intercourse from Visit 1 until the sixth day after the last study visit.
* Willing to abstain from any other vaginal activity and the use of vaginal product other than the study product including tampons, spermicides, lubricants, and douches starting 48 hours before Visit 3 until the sixth day after the last study visit
* Vaginal and cervical anatomy that, in the opinion of the investigator, lends itself to easy colposcopy and genital tract sample collection
* Negative urine pregnancy test
* P4 ≥3 ng/ml
* Willing to give voluntary consent, sign an informed consent form and comply with study procedures as required by the protocol

Exclusion Criteria:

* History of hysterectomy
* Currently pregnant or within two calendar months from the last pregnancy outcome. Note: If recently pregnant must have had at least two spontaneous menses since pregnancy outcome.
* Use of any hormonal contraceptive method in the last 3 months (oral, transdermal, transvaginal, implant, or hormonal intrauterine contraceptive device)
* Injection of Depo-Provera in the last 10 months
* Use of copper intrauterine device (IUD) after Visit 1
* Currently breastfeeding or having breastfed an infant in the last two months, or planning to breastfeed during the course of the study
* History of sensitivity/allergy to any component of: TFV 1% gel, topical anesthetic, or allergy to both silver nitrate and Monsel's solution.
* Contraindication to LNG
* In the last six months, diagnosed with or treated for any sexually transmitted infection (STI) or pelvic inflammatory disease. Note: Women with a history of genital herpes or condylomata who have been asymptomatic for at least six months may be considered for eligibility.
* Nugent score greater than or equal to 7 or symptomatic bacterial vaginosis (BV) as defined by Amsel's criteria
* Positive test for Trichomonas vaginalis, Neisseria gonorrhea (GC), Chlamydia trachomatis (CT), HIV, or Hepatitis B surface antigen (HBsAg)
* Known bleeding disorder that could lead to prolonged or continuous bleeding with biopsy
* Chronic or acute vulvar or vaginal symptoms (pain, irritation, spotting, etc.)
* Known current drug or alcohol abuse which could impact study compliance
* Grade 2 or higher laboratory abnormality, per the August 2009 update of the Division of AIDS, National Institute of Allergy and Infectious Disease (DAIDS) Table for Grading the Severity of Adverse Events, or clinically significant laboratory abnormality as determined by the clinician
* Systemic use in the last two weeks or anticipated use during the study of any of the following: corticosteroids, antibiotics, anticoagulants or other drugs known to prolong bleeding and/or clotting, antifungals, antivirals (e.g., acyclovir or valacyclovir) or antiretrovirals (e.g., Viread, Atripla®, Emtriva®, Complera®). Note: Participants should avoid non-steroidal anti-inflammatory drugs (NSAIDs) except for treatment of dysmenorrhea during menses. Participants may use Tylenol® on an as-needed but not daily basis during the study
* Participation in any other investigational trial (device, drug, or vaginal trial) within the last 30 days or planned participation in any other investigational trial during the study
* History of gynecological procedures (including genital piercing) on the external genitalia, vagina or cervix within the last 14 days
* Abnormal finding on laboratory or physical examination or a social or medical condition which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events | IVR Day 1, 2, ~8, ~16-18; 24 hours and 1-2 weeks post-IVR insertion and 1-2 weeks after IVR removal
  Number of treatment-emergent adverse events
Systemic laboratory tests | Baseline and IVR Day ~16-18
  Changes in Systemic laboratory tests
Cervicovaginal ulcerations, abrasions, edema, and other findings | Baseline, IVR Day 2, ~8 and ~16-18
  Development of cervicovaginal ulcerations, abrasions, edema, and other findings as assessed by naked eye and colposcopic visualization of the cervicovaginal epithelium
Soluble markers of innate mucosal immunity and inflammatory response in cervicovaginal lavage (CVL) fluid | Baseline and IVR Day ~16-18
  Changes in soluble markers of innate mucosal immunity and inflammatory response in CVL fluid
HIV-1 target immune cell phenotype and HIV-1 activation/proliferation marker in cervicovaginal tissue (biopsy) | Baseline and IVR Day ~16-18
  Changes in HIV-1 target immune cell phenotype and HIV-1 activation/proliferation marker in cervicovaginal tissue (biopsy)
Microflora (semi-quantitative vaginal culture and/or unculturable bacteria) | Baseline and IVR Day ~16-18
  Changes microflora (semi-quantitative vaginal culture and/or unculturable bacteria)
Vaginal pH | Baseline and IVR Day ~16-18
  Changes in vaginal pH
Nugent Score | Baseline and IVR Day ~16-18
  Changes in Nugent Score

SECONDARY OUTCOMES:
TFV concentrations in plasma | Baseline; 1, 2, 4 and 8 hrs post-IVR insertion; IVR Day 2, ~8, ~16-18; 24 hours post-IVR removal
  TFV concentrations in plasma
TFV concentrations in cervicovaginal fluid (aspirate and swab) | 1, 2, 4 or 8 hours post-IVR insertion (randomized time point); IVR Day 2, ~8, ~16-18; 24 hours post-IVR removal
  TFV concentrations in cervicovaginal fluid (aspirate and swab)
TFV concentrations in genital tissue (biopsy) | IVR Day 2, ~16-18; 24 or 72 hours post-IVR removal (randomized time point)
  TFV concentrations in genital tissue (biopsy)
Tenofovir diphosphate (TFV-DP) concentrations in peripheral blood mononuclear cells (PBMCs) | IVR Day ~16-18
  TFV-DP concentrations in PBMCs
TFV-DP concentrations in genital tissue (biopsy) | IVR Day 2, ~16-18; 24 or 72 hours post-IVR removal (randomized time point)
  TFV-DP concentrations in genital tissue (biopsy)
LNG concentration in blood (including SHBG) | Baseline; 1, 2, 4 and 8 hrs post-IVR insertion; IVR Day 2, ~8, ~16-18; 24 hours post-IVR removal
  LNG concentration in blood (including SHBG)
LNG concentration in vaginal secretions (swabs) | Baseline; IVR Day~8
  LNG concentration in vaginal secretions (swabs)
LNG concentration in cervical mucus | IVR Day ~8, ~16-18; 24 hours post-IVR removal
  LNG concentration in cervical mucus
Weight of returned IVRs | IVR Day ~16-18 (post-removal)
  Weight of returned IVRs
Amount of drug remaining in returned IVRs | IVR Day ~16-18 (post-removal)
  Amount of drug remaining in returned IVRs

OTHER OUTCOMES:
Cervical mucus assessment and sperm migration on the Simplified Slide test | IVR Day ~8
  Surrogates of contraceptive efficacy - Cervical mucus assessment
Ovulation by P4 | IVR Day ~16-18
  Surrogates of contraceptive efficacy - Ovulation by P4
Follicular development by serum estradiol concentration | IVR Day ~8, ~16-18
  Surrogates of contraceptive efficacy - Follicular development by serum estradiol concentration
Acceptability of IVR | IVR Day ~16-18 (post-removal)
  Acceptability of IVR as measured by a composite of the following factors: Discontinuations, Expulsions, Removals, Visible changes (such as discoloration) as documented on photographs of returned IVRs, Responses to key questions on acceptability questionnaire
Pharmacodynamics | Baseline, IVR Day ~16-18
  Pharmacodynamics - Anti-herpes simplex virus (HSV)-2 and Anti-HIV-1 activities in the CVL. Anti-HIV and anti-HSV activity as a percent of anti-HIV and anti-HSV activity before exposure to test product
Pharmacodynamics | Baseline, IVR Day ~16-18
  TFV anti-HIV efficacy in cervicovaginal tissues. Comparison of cervicovaginal tissue permissiveness to ex vivo infection with HIV-1 BaL between the control cycle and treatment cycle.
Pharmacodynamic surrogates of LNG in endometrium | Baseline, IVR Day ~16-18
  Findings on endometrial biopsy: Histology, Markers of endometrial function
Endometrial thickness | Baseline, IVR Day ~16-18
  Endometrial thickness as assessed by transvaginal ultrasound
Cervicovaginal epithelial histology and epithelial integrity in cervicovaginal tissue (biopsy) | Baseline, IVR Day ~16-18
  Cervicovaginal epithelial histology (thickness and number of cell layers) and epithelial integrity, as measured immuno-histochemistry (IHC) of epithelial junction proteins in cervicovaginal tissue (biopsy)
Markers of mucosal alteration and inflammation (e.g., expression of COX-2) in cervicovaginal and endometrial tissue | Baseline, IVR Day ~16-18
  Markers of mucosal alteration and inflammation (e.g., expression of COX-2) in cervicovaginal and endometrial tissue
Microbial growth on swabs obtained from returned IVRs and microbial levels in returned IVRs | IVR Day ~16-18 (post-removal)
  Microbial growth on swabs obtained from returned IVRs and microbial levels in returned IVRs
Level of association of TFV levels between less-invasive swabs and the more invasive biopsies, and possibly between swabs and aspirates | IVR Day 2, ~16-18; 24 hours post-IVR removal
  Level of association of TFV levels between less-invasive swabs and the more invasive biopsies, and possibly between swabs and aspirates
Characterization of returned IVRs for physicochemical properties and potential chemical and/or biological measures of adherence | IVR Day ~16-18 (post-removal)
  Characterization of returned IVRs for physicochemical properties and potential chemical and/or biological measures of adherence

CONTACTS AND LOCATIONS:
Overall Officials: Jill Schwartz, MD, Study Chair — CONRAD; Chris Mauck, MD, Study Director — CONRAD
Locations (2):
- Eastern Virginia Medical School, Norfolk, Virginia, United States
- Profamilia, Santo Domingo, Dominican Republic, Dominican Republic

REFERENCES:
- [Derived] Thurman AR, Schwartz JL, Ravel J, Gajer P, Marzinke MA, Yousefieh N, Anderson SM, Doncel GF. Vaginal microbiota and mucosal pharmacokinetics of tenofovir in healthy women using tenofovir and tenofovir/levonorgestrel vaginal rings. PLoS One. 2019 May 20;14(5):e0217229. doi: 10.1371/journal.pone.0217229. eCollection 2019. PMID 31107913
- [Derived] Thurman AR, Schwartz JL, Brache V, Clark MR, McCormick T, Chandra N, Marzinke MA, Stanczyk FZ, Dezzutti CS, Hillier SL, Herold BC, Fichorova R, Asin SN, Rollenhagen C, Weiner D, Kiser P, Doncel GF. Randomized, placebo controlled phase I trial of safety, pharmacokinetics, pharmacodynamics and acceptability of tenofovir and tenofovir plus levonorgestrel vaginal rings in women. PLoS One. 2018 Jun 28;13(6):e0199778. doi: 10.1371/journal.pone.0199778. eCollection 2018. PMID 29953547